CLINICAL TRIAL: NCT06753916
Title: Multicenter Clinical Trial to Evaluate the Safety and Efficacy of Ex Vivo Corneal Cross-linking of Donor Corneal Tissue Used for Vascularized High-risk Keratoplasty
Brief Title: ExCrossV Multi Site Trial for Vascularized High Risk Keratoplasty
Acronym: ExCrossV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Joseph B. Ciolino, MD, Associate Professor of Ophthalmology, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023P002687
Record Dates: First submitted 2024-09-19; First posted 2024-12-31 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Corneal Transplant Failure
Keywords: Keratoplasty; Cross Linking
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants Receiving Treated Cross Linked Corneal Tissue (Experimental): Participants in this group will receive tissue that has been treated with 0.1% riboflavin (Vitamin B2) and 20% dextran (Photrexa® viscous and Photrexa®) with UV light treatment. Participants will be monitored over a period of 24 months.
  Interventions: Procedure: Corneal Donor Tissue with Cross Linking
- Participants Receiving Untreated Cross Linked Corneal Tissue (Placebo Comparator): Participants in this group will receive tissue that has has not been treated with 0.1% riboflavin (Vitamin B2) and 20% dextran (Photrexa® viscous and Photrexa®) without UV light treatment. Participants will be monitored over a period of 24 months.
  Interventions: Procedure: Corneal Donor Tissue without Cross Linking

INTERVENTIONS:
Procedure: Corneal Donor Tissue with Cross Linking — Participants are transplanted with corneal donor tissue that has been treated with 0.1% riboflavin (Vitamin B2) and 20% dextran (Photrexa® Viscous & Photrexa®) with UV light treatment.
  Other Names: Treatment
  Arms: Participants Receiving Treated Cross Linked Corneal Tissue
Procedure: Corneal Donor Tissue without Cross Linking — Participants are transplanted with corneal donor tissue that has not been treated with the UV light and the 0.1% riboflavin (Vitamin B2) and 20% dextran (Photrexa® Viscous & Photrexa®) without UV light treatment, this is the control group.
  Other Names: Control
  Arms: Participants Receiving Untreated Cross Linked Corneal Tissue

SUMMARY:
The main objective of this study is to determine the safety of Ex Vivo Cross Linking (CXL) of donor corneal tissue in participants who have undergone high-risk penetrating keratoplasty.

DETAILED DESCRIPTION:
This is a randomized, double-masked, multi site clinical trial to determine the safety of Ex Vivo CXL of donor corneal tissue in 96 participants who have undergone high-risk penetrating keratoplasty.

Participants will be randomized to receive either a corneal tissue that has been untreated vs. a corneal tissue that has been treated with Photrexa® Viscous & Photrexa® and UV light. The tissue will be prepared by a Corneal Tissue Bank under Current-Good-Tissue-Practice (CGTP) and delivered to the respective institutions for transplantation. Participants will be monitored up to 24 months post-transplantation to assess for adverse events of the randomized tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Willing and able to provide written informed consent
* Willing and able to comply with study assessments for the full duration of the study
* Patients undergoing high-risk penetrating keratoplasty, defined as corneal neovascularization (NV) in 1 or more quadrants ≥2 mm from the limbus or extension of corneal NV to the graft-host junction in a previously failed graft
* Superficial vessels are defined as those within the anterior one-third of the cornea and deep vessels within the posterior two-thirds of the cornea (i.e., deep stroma).

Superficial CNV involving ≤2 quadrants (equivalent to ≤6 clock hours) without deep CNV are classified as mild. CNV with >2 quadrants of superficial vessels (>6 clock hours) or 1 quadrant of deep vessels (>3 clock hours) as severe (36).

Exclusion Criteria:

* History of Stevens-Johnson syndrome or ocular pemphigoid
* Ocular or periocular malignancy
* Non-healing epithelial defect of at least 0.5x0.5 mm in host corneal bed lasting ≥6 weeks preoperatively
* Uncontrolled glaucoma
* Change in topical corticosteroid regimen within 14 days of transplantation
* Use of systemic immunosuppressive for indication other than corneal graft rejection
* Participation in another simultaneous medical investigation or trial
* Pregnancy (positive pregnancy test) or lactating
* Pre-menopausal women not using adequate contraception (Reliable intrauterine devices, hormonal contraception or a spermicide in combination with a barrier method)
* Ocular infection within 30 days prior to study entry.
* Presence of anterior chamber intraocular lens
* Active uveitis within 90 days prior to the study entry.
* No ocular surgery or procedure within 90 days prior to the study entry or concomitant to the study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Determining the Primary Safety of Corneal Cross Linking | 24 Months
  The occurrence of adverse events throughout study including:
  1. Ocular Safety per the incidences and severity of ocular adverse events during the study based on ophthalmic examination and participants' self-report.
  2. Short Term Safety Events (Post Surgery < 1 Month)
     * Post-Op Microbial Keratitis
     * Acute Rejection (Epithelial, Endothelial, Sub epithelial, or Mixed)
  3. Long Term Safety Events (Post Surgery > 1 Month)
     * Rejection (Epithelial, Endothelial, or Mixed)
     * Graft Failure
     * Ulcerative Keratitis
     * Persistent Epithelial Defect lasting more than 6 Weeks

SECONDARY OUTCOMES:
Measure of the Frequency of Graft Failures though Corneal Cross Linking | 24 Months
  To determine the efficacy of using cross linked tissue for the indicated keratoplasty for the prevention of corneal graft rejection and corneal neovascularization, by measuring the frequency of primary graft failures over 24 months.
Measure of Time from Surgery to Overall Graft Failure for Corneal Cross Linking over 24 Months | 24 Months
  The efficacy of using cross linked tissue for the indicated keratoplasty for the prevention of corneal graft rejection and corneal neovascularization, by measuring the time from surgery to overall graft failure (regardless of cause).
Measure of Time from Surgery to Graft Rejection for Corneal Cross Linking over 24 Months | 24 Months
  The efficacy of using cross linked tissue for the indicated keratoplasty for the prevention of corneal graft rejection and corneal neovascularization, by measuring the occurrence of any rejection episode. (Epithelial, Endothelia, Sub Epithelial, or Mixed) determined as either definite rejection, probably rejection, and possible rejection, from the time of surgery over 24 months.
Measure of the Efficacy of Corneal Cross Linking Through Image Review | 24 Months
  The efficacy of using cross linked tissue for the indicated keratoplasty for the prevention of corneal graft rejection and corneal neovascularization.
  1. Corneal Neovascularization (CNV) measured and analyzed from slit-lamp photography.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ciolino, MD, Principal Investigator — Massachusetts Eye and Ear
Locations (12):
- United States (12):
  - University of California Irvine - Gavin Herbert Eye Institute, Irvine, California
  - The University of California Los Angeles - Doris Stein Eye Research Center, Los Angeles, California
  - University of California San Francisco - Wayne and Gladys Valley Center for Vision, San Francisco, California
  - University of Miami - Bascom Palmer Eye Institute, Miami, Florida
  - Price Vision Group, Indianapolis, Indiana
  - Kansas City Eye Clinic, Overland Park, Kansas
  - Mid-Atlantic Cornea Consultant, Towson, Maryland
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - University of Michigan - Kellogg Eye Center, Ann Arbor, Michigan
  - Wake Forest Baptist Eye Center, Bermuda Run, North Carolina
  - Duke University - Duke Eye Center, Durham, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio